CLINICAL TRIAL: NCT02319993
Title: Traditional Chinese Medicine Suan Tsao Jen Tang and Tian-Wang-Bu-Xin Dan in Patients With Primary Insomnia. A Multi-center Clinical Trial
Brief Title: Traditional Chinese Medicine Suan Tsao Jen Tang and Tian-Wang-Bu-Xin Dan in Patients With Primary Insomnia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, GCRC, Chief, Department of Critical Care Medicine and Division of Pulmonary Medicine, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSH-CMCTC-101-001
Record Dates: First submitted 2014-12-14; First posted 2014-12-19 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Insomnia
Keywords: Suan-Zao-Ren Tang; Tian-wang-bu-xin-dan; Traditional Chinese Medicine; Herbs; Quality of life
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TIAN WANG BU XIN DAN (Experimental): Drug:TIAN WANG BU XIN DAN CONCENRATED GRANULES "CHUANG SONG ZONG"
  Interventions: Drug: TIAN WANG BU XIN DAN
- Suan Tzao Ren Tang (Experimental): Drug:Suan Tzao Ren Tang Granula Subtilae "CHUANG SONG ZONG"
  Interventions: Drug: Suan Tzao Ren Tang
- Placebo (Placebo Comparator): Drug:1/10 TIAN WANG BU XIN DAN
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TIAN WANG BU XIN DAN — assigned to TWBXD (n =48) and were instructed to take 6 gm 2 times per day of TWBXD for a period of 4 weeks.
  Other Names: TWBXD
  Arms: TIAN WANG BU XIN DAN
Drug: Suan Tzao Ren Tang — assigned to SZRT (n = 48) and were instructed to take 6 gm 2 times per day of SZRT for a period of 4 weeks.
  Other Names: STRT
  Arms: Suan Tzao Ren Tang
Drug: Placebo — 1/10 TIAN WANG BU XIN DAN assigned to placebo (n =32) and were instructed to take 6 gm 2 times per day of placebo for a period of 4 weeks.
  Other Names: P
  Arms: Placebo

SUMMARY:
keywords： Traditional Chinese Medicine, Herbs, Clinical trial, Insomnia, Quality of life, Suan-Zao-Ren Tang, Tian-wang-bu-xin-dan

DETAILED DESCRIPTION:
Title： Traditional Chinese Medicine Suan Tsao Jen Tang and Tian-Wang-Bu-Xin Dan in patients with primary insomnia. A multi-center, double blind, placebo controlled clinical trial.

(First year of two-years' project)

Design:

Randomized, placebo-controlled trial comprising 3 arms: SZRT, placebo, TWBXD.

Setting:

The Chung Shan Medical University Affiliated Hospital and the Taipei City Hospital.

Methods:

A total of 128 subjects 20-80 years of age with a history of insomnia at least 1 month were recruited randomly assigned to SZRT (n = 48), placebo (n =32), TWBXD (n =48) and were instructed to take 6 gm 2 times per day of SZRT, TWBXD or placebo for a period of 4 weeks. The primary outcome measures were the mean component scores of the Pittsburgh Sleep Quality Index (PSQI). Secondary outcome parameter were the global score on the World Health Organization Quality of Life questionnaire - Taiwan brief version, drugs consumption counts, sleep diary and safety profiles by structures questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia disorders in patients 20-80 years of age, the Pittsburgh Sleep Assessment Scale (PSQI)> 6 points.
* No insomnia caused by other diseases. For example: mental illness (depression, etc.), sleep apnea, heart disease (acute myocardial infarction, heart rate is not the whole), hypertension, diabetes, cancer and so on.
* There are more than a week (including) three times to be more than 30 minutes to fall asleep and sleep less than six hours, there is a continuous months.
* Test subjects had to really understand the nature of this study, and participants signed consent.

Exclusion Criteria:

* Before participating in this study, three months, had a major accident or wheel graveyard shift or jet lag problems (such as a long flight).
* Any insomnia caused by other diseases. For example: mental illness (depression, etc.), sleep apnea, heart disease (acute myocardial infarction), poorly controlled hypertension (> 140 / 90mmHg), poorly controlled diabetes (HbA1C> 7%), cancer, digestive ulcers (undergoing treatment).
* 2 weeks into the experiment of taking melatonin or melatonin agonist, acetylcholine, glutamate, serotonin, norepinephrine, GABA, histamine, adenosine, prostaglandins and other drugs.
* If patients sleep disorders arise from nighttime urinary frequency. Pregnant or breastfeeding person.
* Patients unable to read and fill out the questionnaire by themselves this study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 4 weeks

SECONDARY OUTCOMES:
World Health Organization Quality of Life questionnaire | 4 weeks